CLINICAL TRIAL: NCT01069549
Title: Study of the Association of AGTR1 and ACACB Gene Polymorphism and Susceptibility of Diabetic Nephropathy in North Indian Type 2 Diabetic Patients
Brief Title: Association of AGTR1 and ACACB Gene Polymorphism and Diabetic Nephropathy in Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Anil Bhansali, prof and head, Post Graduate Institute of Medical Education and Research, Chandigarh
Organization: PIMERIndia (Unknown)
Other Study IDs: AT1RGPT2DM
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2015-10-26 (Estimated); Status verified 2015-10

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Type 2 Diabetes Mellitus; Diabetic Nephropathy; Angiotensin II type 1 receptor gene polymorphism; Acetyl coA carboxylase beta gene polymorphism.
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetic Nephropathies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 4 ml of whole blood sample.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- subjects with diabetic nephropathy.: Subjects with Type 2 Diabetes. Duration of diabetes should be more than or equal to 5 years. Age between 30 and 85 years. Diabetic nephropathy as defined by ADA.
  Subject must be of north Indian origin.
  Type 1 diabetes and kidney disease other than diabetes nephropathy are excluded form the study.
- Subjects without Diabetic nephropathy.: This group of subject with similar characteristics as group 1 without any evidence of nephropathy.

SUMMARY:
India is the "Diabetes Capital of the World" with 41 million Indians having diabetes, with every fifth diabetic in the world being an Indian and type 2 Diabetes Mellitus (T2DM) constitutes the major chunk of diabetes. One of the most severe complications of diabetes is the development of diabetic nephropathy. Diabetic nephropathy (DN) is the leading cause of end-stage renal disease (ESRD) worldwide. There are many identifiable risk factors of diabetic nephropathy like hyperglycemia, hyperlipidemia, hypertension, and proteinuria, the genetic factor is the main among all. Long-term observational studies show that nearly 30-35% of type 2 diabetic patients develop nephropathy, irrespective of glycemic control. The regional variation in diabetes prevalence and in the proclivity for diabetes induced renal disease; along with reports of familial clustering of nephropathy suggest a possible genetic basis. The renin-angiotensin system (RAS) has been strongly implicated in the pathogenesis of progressive renal diseases. In addition, the blockage of angiotensin II with either ACE inhibitor or an angiotensin type-I receptor antagonist has been found to prevent or delay the progression of renal injury associated with diabetes 5 and now these drugs are first-choice drugs for the treatment of diabetic subjects with hypertension. The genes encoding the renin-angiotensin system (RAS), such as angiotensin-converting enzyme (ACE), angiotensinogen (AGT) and angiotensin II receptor type 1 (AGTR1), have been reported to be the most probable candidate genes for diabetic nephropathy. As there is no data available for AGTR1 polymorphism and DN in the north Indian T2DM, its out attempt to fill the scientific gap.

ELIGIBILITY:
Group:-1: Patients with diabetic nephropathy

Inclusion criteria:

* Type 2 Diabetes and duration of more than or equal to 5 years.
* Age between 30 to 85 years.
* Presence of both albuminuria and retinopathy.

Exclusion criteria:

* Patients with diagnosis of type 1 diabetes
* Any known nondiabetic renal disease.
* Patients who had a MI or had undergone CABG within 3 month.
* Patients who had a CVA or had undergone PTCA in the previous 3 months.
* Patients who had had a transient ischemic attack within the previous 3 months.
* Patients who had any history of heart failure before enrollment.
* Patients with UTI.
* Pregnant patient.

Group:-2: Patients without diabetic nephropathy Same characteristic as group 1 but no evidence of diabetic nephropathy.

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study Population for Group 1 and Group-2 (Subjects with diabetic nephropathy and without nephropathy respectively)will be recruited from the diabetic Out Patient and in patient services of Postgraduate Institute of Medical Education & Research and Nehru hospital, Chandigarh. Only North Indian Ethnic subjects will be recruited.
Sampling Method: Non-Probability Sample
Enrollment: 476 (Actual)
Dates: Start 2009-11; Primary Completion 2011-04 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: anil Bhansali, DM, Study Chair — Postgradute Institute of Medical Education & Research
Locations (1):
- Postgraduate Institute of Medical Education & Research, Chandigarh, Chandigarh, India